CLINICAL TRIAL: NCT06119477
Title: Comparison of Three Techniques in Bioceramic Apexification Procedure for Necrotic Immature Incisors: A Randomized Clinical Trial
Brief Title: Three Techniques in Bioceramic Apexification for Necrotic Immature Incisors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Pedo-06-2023
Record Dates: First submitted 2023-10-22; First posted 2023-11-07 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Immature Teeth; Periapical Lesion
Keywords: post-operative pain; periapical lesion healing; bioceramic apexification
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bioceramic Putty Apical Plugs (Experimental): The Bioceramic Putty will be inserted in the apical 4 mm of the canal using the modified cannula and adapted to the canal walls with a hand plugger.
  Interventions: Other: Bioceramic Putty Apical Plugs
- Single Cone Gutta-percha with Bioceramic Sealer (Experimental): A large sized (#80 - #120, and a taper of 2%) gutta-percha cone (GC) will be inserted, measuring according to the width of the canal, to the working length, then the immature canal will be gently filled with Bioceramic sealer and the GC.
  Interventions: Other: Single Cone Gutta-percha with Bioceramic Sealer
- Combination of Bioceramic Putty and Sealer (Experimental): The immature canal will be gently filled with Bioceramic sealer and then 3 to 5 small balls of BP will be inserted into the canal orifice and gently plugged with hand pluggers.
  Interventions: Other: Combination of Bioceramic Putty and Sealer

INTERVENTIONS:
Other: Bioceramic Putty Apical Plugs — Under local anesthesia and rubber dam isolation, the canal orifice will be prepared gently. The working length and apex diameter value will be recorded as a reference. Afterward, shaping and debridement the root canals will be achieved by gentle instrumentation. The canal will be irrigated copiously with NaOCl, then dried, and filled with Ca(OH)2 dressing. Afterward, the incisor will be temporarily restored. After 14 days the temporary filling and Ca(OH)2 will be removed. Afterward, canals will be irrigated with NaOCl and EDTA and dried. The Bioceramic Putty will be inserted in the apical 4 mm of the canal using the modified cannula and adapted to the canal walls with a hand plugger. The correct placement and thickness of the apical plug will be verified with a periapical radiograph. Afterward, the remainder of the root canal will be filled with gutta-percha with sealer. Finally, a suitable immediate final restoration was made for each case individually.
  Arms: Bioceramic Putty Apical Plugs
Other: Single Cone Gutta-percha with Bioceramic Sealer — Under local anesthesia and rubber dam isolation, the canal orifice will be prepared gently. The working length and apex diameter value will be recorded as a reference. Afterward, shaping and debridement the root canals will be achieved by gentle instrumentation. The canal will be irrigated copiously with NaOCl, dried, filled with Ca(OH)2 dressing and temporarily restored. After 14 days the temporary filling and Ca(OH)2 will be removed. Afterward, canals will be irrigated with NaOCl and EDTA and dried. A large sized gutta-percha cone (GC) will be inserted to the working length, The GC was ensured to make tag-back with the apical third of the immature canal and confirmed with a periapical radiograph. Then the immature canal will be gently filled with Bioceramic sealer and the GC will be placed again and another apical radiograph will be taken to confirm that the canal was properly filled. Finally, a suitable immediate final restoration was made for each case individually.
  Arms: Single Cone Gutta-percha with Bioceramic Sealer
Other: Combination of Bioceramic Putty and Sealer — Under local anesthesia and rubber dam isolation, the canal orifice will be prepared gently. The working length and apex diameter value will be recorded as a reference. Afterward, shaping and debridement the root canals will be achieved by gentle instrumentation. The canal will be irrigated copiously with NaOCl, dried, filled with Ca(OH)2 dressing and temporarily restored. After 14 days the temporary filling and Ca(OH)2 will be removed. Afterward, canals will be irrigated with NaOCl and EDTA and dried.
  The immature canal will be gently filled with Bioceramic sealer and then 3 to 5 small balls of BP (diameter of 1 mm) will be inserted into the canal orifice and gently plugged with hand pluggers. Afterward, an apical radiograph will be taken to confirm that the canal was properly filled without gaps and voids. Finally, a suitable immediate final restoration was made for each case individually.
  Arms: Combination of Bioceramic Putty and Sealer

SUMMARY:
The goal of this randomized clinical trial is to find the most effective Bioceramic-based apexification procedures in children with immature necrotic maxillary incisors. The main questions they aims to answer are:

* What is the best Bioceramic apexification technique regarding the post-operative pain and the periapical healing ?
* What is the best Bioceramic apexification technique regarding the bioceramics extrusion and the required time ? Participants will under gone Bioceramic apexification procedures which root canal preparing, disinfecting, filling, and restoring. Then, the patient will asked to come to follow-up appointments for clinical and radiological evaluations If there is a comparison group: Researchers will compare Bioceramic Putty Apical Plugs, Single Cone Gutta-percha with Bioceramic Sealer, and Combination of Bioceramic putty and sealer technique to find the best effective technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more maxillary incisors with an open apex root (defined as root which root canal size equal or larger than #80 K-file) and presented with pulp necrosis and radiographic evidence of chronic apical periodontitis and periapical radiolucency greater than 3 mm.

Exclusion Criteria:

* Children with systemic diseases that compromised their general immune status.
* Uncooperative (definitely negative on the Frankl's behavioral scale).
* unrestorable incisors.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation | 12 months
  Patients of both groups will be recalled after 1, 3, 7, and 14 days of treatment and during radiographical assessment periods (3, 6 and 12 months), where they will be asked to rate their pain on the Wong-Baker Faces Scale, where children will set their pain levels by choosing a face; 0 = No Hurt, 1 = Hurts little bit, 2 = hurts Little more 3 = Hurts even more, 4 = Hurts whole lot, and 5 = Hurts worst. Moreover, the presence of fistula, swelling, and movement will be recorded.
Radiographical assessment | 12 months
  After coronal restoration is completed a control x-ray will be taken. The periapical status will be assessed at the time of obturation-restoration, 3, 6, and 12 months following endodontic treatment. The outcome will be determined according to the Periapical Index scoring system: (1) normal periapical structures (The best); (2) small changes in bone structure; (3) changes in bone structure with some mineral loss; (4) periodontitis with well-defined radiolucent area; (5) severe periodontitis with exacerbating features (The worst).
  The teeth will be evaluated according to healed, healing or unsuccessful as a primary radiographical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Aljabban, Proffesor, Study Director — Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
only with contacting the main researcher

REFERENCES:
- [Background] Tolibah YA, Kouchaji C, Lazkani T, Ahmad IA, Baghdadi ZD. Comparison of MTA versus Biodentine in Apexification Procedure for Nonvital Immature First Permanent Molars: A Randomized Clinical Trial. Children (Basel). 2022 Mar 14;9(3):410. doi: 10.3390/children9030410. PMID 35327782
- [Derived] Alsayed Tolibah Y, Bshara N, Abbara MT, Alhaji M, Aljabban O, Ahmad IA, Baghdadi ZD. Root Development Following Bioceramic Material Application in Immature Permanent Teeth: A Case Series With 24-Month Follow-Up. Case Rep Dent. 2025 Oct 22;2025:1530438. doi: 10.1155/crid/1530438. eCollection 2025. PMID 41169957